CLINICAL TRIAL: NCT03296202
Title: Risk of Morbidity, Mortality and Long-term Monitoring of Antiretroviral Treatment in People Living With HIV: The ANRS CO3 Aquitaine Cohort - AquiVIH-NA
Brief Title: Risk of Morbidity, Mortality and Long-term Monitoring of Antiretroviral Treatment in People Living With HIV
Acronym: AquiVIH-NA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: National Agency for Research on AIDS and Viral Hepatitis (ANRS) (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); French Ministry of Health through the COREVIH Aquitaine (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/04
Record Dates: First submitted 2017-06-23; First posted 2017-09-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections; Antiretroviral Agents
Keywords: HIV; cohort studies; antiretroviral treatment
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV patients: 7200 patients infected with HIV-1

SUMMARY:
HIV infection is now a chronic disease in countries where antiretroviral treatments (ART) are largely available. Long-term follow-up is required to describe and understand the evolution of morbidities and complications as well as new treatments side effects.

The main objective of the cohort is to describe and study the evolution of HIV infection in ART-treated individuals.

DETAILED DESCRIPTION:
The survival of people living with HIV (PLHIV) taking antiretroviral therapy (ART) is now close to what is reported in the general population in northern countries. However, PLHIV experience an increased risk of morbidities that the ANRS CO3 Aquitaine Cohort has largely contributed to describe in the last years. Among contributing factors to this excess of morbidity, immune suppression, immune activation, and exposition to cardiovascular and cancer risk factors as well as ageing represent possible intervention targets. Long-term follow-up is required to describe and understand the evolution of morbidities and complications as well as ART side effects.

Moreover, the global evaluation of health in PLHIV, including psychiatric, neurologic and social determinants and not only biomedical determinants represents one of the public health challenges of the next decade in the field of HIV infection.

The aim of the present study is to study the emerging morbidity occurring during the course of HIV infection in people treated with ART as well as to describe the tolerance and efficacy of new available ART regimens.

The follow-up of patients will be performed according to national guidelines. Demographic, clinical, biological and therapeutic data will be captured at each patient's hospital contact according to a standardized questionnaire.

All events occurring during the course of clinical management will be prospectively registered in the database according to the ICD 10th revision. A biobank will be collected from every consenting PLHIV at inclusion in the cohort and then every two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old.
* Confirmed HIV infection
* Signed informed consent

Exclusion Criteria:

* HIV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with HIV-1 (PLHIV)
Sampling Method: Non-Probability Sample
Enrollment: 7200 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Socio-demographic characteristics of people living with the HIV | Each 12 months from baseline for 4 years (M48)

SECONDARY OUTCOMES:
HIV infection characteristics of people living with the HIV | Each 12 months from baseline for 4 years (M48)
  group of infection, stage of infection, duration since first serology positive, CD4 nadir, last CD4 measurement, CD4 / CD8 ratio
comorbidities of people living with the HIV | Each 12 months from baseline for 4 years (M48)
co-infections of people living with the HIV | Each 12 months from baseline for 4 years (M48)
  Hepatitis B, Hepatitis C, cytomegalovirus infection...
Therapeutics description | Each 12 months from baseline for 4 years (M48)
  naïve / treated status, dosage
virological responses | Each 12 months from baseline for 4 years (M48)

CONTACTS AND LOCATIONS:
Overall Officials: Linda WITTKOP, MD, PhD, Study Chair — ISPED - CHU de Bordeaux; Fabrice BONNET, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (22):
- France (22):
  - service de médecine interne - CH d'Agen, Agen
  - Médecine interne - CH d'Angoulême, Angoulême
  - service de maladies infectieuses - CH de la Côte Basque, Bayonne
  - service de médecine inter et maladies infectieuses - Hopital Saint André, Bordeaux
  - service de médecine interne et maladies infectieuses - Hôpital Saint-André, Bordeaux
  - service de maladies infectieuses et médecine tropicale - Hôpital Pellegrin, Bordeaux
  - Service D'Urgences Pédiatriques, Bordeaux
  - médecine interne - CH de Châtellerault, Châtellerault
  - service de médecine interne et maladies infectieuses - CH de Dax, Dax
  - Médecine Interne - CH de Jonzac, Jonzac
  - service de médecine interne - CH d'Arcachon, La Teste-de-Buch
  - service de médecine interne - CH de Libourne, Libourne
  - service de médecine interne - CH de Mont de Marsan, Mont-de-Marsan
  - service de médecine interne - CH d'Orthez, Orthez
  - service de médecine interne et maladies infectieuses - CH de Pau, Pau
  - service de médecine interne et maladies infectieuses - Groupe hospitalier Sud, Pessac
  - service de médecine interne et maladies infectieuses - CH de Périgueux, Périgueux
  - Médecine interne et Maladies Infectieuses - CHU de Poitiers, Poitiers
  - Médecine interne - CH de Royan, Royan
  - Médecine Interne - CH de Saint-Jean-D'Angely, Saint-Jean-d'Angély
  - Médecine Interne - CH de Saintonge, Saintes
  - service de maladies infecteieuses - CH Saint-Cyr, Villeneuve-sur-Lot

REFERENCES:
- [Derived] Devos S, Bonnet F, Hessamfar M, Neau D, Vareil MO, Leleux O, Cazanave C, Rouanes N, Duffau P, Lazaro E, Dabis F, Wittkop L, Barger D; ANRS CO3-AQUIVIH-NA-QuAliV. Tobacco, alcohol, cannabis, and illicit drug use and their association with CD4/CD8 cell count ratio in people with controlled HIV: a cross-sectional study (ANRS CO3 AQUIVIH-NA-QuAliV). BMC Infect Dis. 2023 Jan 9;23(1):16. doi: 10.1186/s12879-022-07963-6. PMID 36624391
- [Derived] Barger D, Hessamfar M, Neau D, Vareil MO, Lazaro E, Duffau P, Rouanes N, Leleux O, Le Marec F, Erramouspe M, Wittkop L, Dabis F, Bonnet F. Assessing the psychometric properties of the French WHOQOL-HIV BREF within the ANRS CO3 Aquitaine Cohort's QuAliV ancillary study. Health Qual Life Outcomes. 2020 Jul 10;18(1):220. doi: 10.1186/s12955-020-01451-8. PMID 32650781
- [Derived] Barger D, Leleux O, Conte V, Sapparrart V, Gapillout M, Crespel I, Erramouspe M, Delveaux S, Wittkop L, Dabis F, Bonnet F. Web-Based Module for the Collection of Electronic Patient-Reported Outcomes in People Living With HIV in Nouvelle Aquitaine, France: Usability Evaluation. JMIR Form Res. 2019 Dec 18;3(4):e15013. doi: 10.2196/15013. PMID 31850847
- [Derived] Barger D, Leleux O, Conte V, Sapparrart V, Gapillout M, Crespel I, Erramouspe M, Delveaux S, Dabis F, Bonnet F. Integrating Electronic Patient-Reported Outcome Measures into Routine HIV Care and the ANRS CO3 Aquitaine Cohort's Data Capture and Visualization System (QuAliV): Protocol for a Formative Research Study. JMIR Res Protoc. 2018 Jun 7;7(6):e147. doi: 10.2196/resprot.9439. PMID 29880467